CLINICAL TRIAL: NCT03119701
Title: A Randomised, Parallel Group 2:1 Comparison of the Efficacy and Safety of FP-1201-lyo (Interferon Beta-1a) and Placebo in the Prevention of Multi-Organ Failure on Patients Surviving Open Surgery for a Ruptured Abdominal Aortic Aneurysm
Brief Title: Efficacy and Safety of FP-1201-lyo (Interferon Beta-1a) in Prevention of Multi-Organ Failure on Patients After Open Surgery for a RAAA
Acronym: INFORAAA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: IDMC recommendation. Unexpectedly high use of concomitant corticosteroid treatment.
Sponsor: Faron Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FP1CLI006; 2014-000899-25 (EudraCT Number)
Record Dates: First submitted 2017-03-03; First posted 2017-04-19 (Actual); Results first posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2020-12

CONDITIONS: Preventive Medicine; Multi Organ Failure
Keywords: Patients Surviving Open Surgery; Ruptured Abdominal Aortic Aneurysm
MeSH Terms: conditions — Multiple Organ Failure | interventions — Interferon beta-1a; Drugs, Investigational

STUDY DESIGN:
Intervention Model Description: Multicentre, randomised, double-blinded, Phase II, parallel group comparison study of the efficacy and safety of FP-1201-lyo compared to placebo in patients surviving emergency open surgery for an infra-renal ruptured abdominal aortic aneurysm.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FP-1201-lyo 10 µg (Experimental): FP-12-lyo 10 µg (Interferon Beta-1a) will be administered once daily as an intravenous bolus injection for 6 days.
  Investigational product is lyophilisate for solution for injection which will be reconstituted in water for injection.
  Interventions: Drug: Interferon Beta-1A
- FP-1201-lyo Placebo (Placebo Comparator): FP-1201-lyo Placebo will be administered once daily as an intravenous bolus injection for 6 days.
  Investigational placebo is lyophilisate for solution for injection which will be reconstituted in water for injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Interferon Beta-1A — Lyophilisate for solution for injection.
  Other Names: FP-1201-lyo; ATC code L03AB07
  Arms: FP-1201-lyo 10 µg
Drug: Placebo — Lyophilisate for solution for injection as placebo.
  Other Names: Placebo for investigational drug
  Arms: FP-1201-lyo Placebo

SUMMARY:
A study to assess effectiveness and safety of a drug FP-1201-lyo (Recombinant Human Interferon Beta-1a) in the Prevention of Multi-Organ Failure on patients after Open Surgery for a Ruptured Abdominal Aortic Aneurysm

DETAILED DESCRIPTION:
This trial is multicentre, randomised, double-blinded, Phase II, parallel group comparison study of the efficacy and safety of FP-1201-lyo compared to placebo in patients surviving emergency open surgery for an infra-renal ruptured abdominal aortic aneurysm. Investigational medicinal product will be administered as post-surgical preventive treatment either 10µg FP-1201-lyo or placebo. Treatment will be administered daily every 24 hrs for 6 days. The first dose will be given after successful surgery at the point when the patient arrives to the Intensive Care Unit (ICU).

Both treatment groups will receive standard supportive care.

Aim is randomise and initiate treatment of 152 patients. For the final analysis, a minimum of 129 evaluable patients will be required.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion into this study, each patient must fulfil the following inclusion criteria during screening and prior to the first dose of study medication being administered on D0 (criteria 1 or 2 and all 3, 4 and 5):

1. Patients (male or female) presenting with a ruptured abdominal aortic aneurysm (RAAA) diagnosed by ultrasound or CT-scan in the emergency room

   * all forms of infrarenal RAAAs with or without coexisting iliac aneurysms are included or
2. Patients (male or female) presenting with symptoms of RAAA known to have an infrarenal AAA and proceeding straight to open repair without radiological assessment and confirmed rupture (=retroperitoneal haematoma) in operation

   and
3. Aneurysma repair must be infra-renal, i.e. the proximal anastomosis must be below the renal arteries and the renal arteries have to stay intact. Temporary above the renal clamping can be used for a maximum of 30 minutes (total clamping time)

   and
4. Patients providing informed consent

   and
5. Age of 18 years or higher

Exclusion Criteria:

To be eligible for inclusion into this study, each patient must not meet any of the following exclusion criteria during screening or prior to the first dose of study medication being administered:

1. Moribund patient not eligible for treatment in ICU or expected to survive surgery
2. Markedly short life expectancy, e.g. advanced malignant disease
3. Current participation in another experimental treatment protocol
4. Significant congestive heart failure, defined as New York Heart Association (NYHA) class IV
5. Current treatment with Interferon (IFN) alpha or IFN beta
6. Dialysis therapy for chronic renal failure
7. Irreversible shock from haemorrhage
8. Unconsciousness or inability to give consent
9. Ruptured Endovascular Aortic Repair (rEVAR) first (prior attempt for endovascular aortic repair for the current rupture)
10. Diagnosed cirrhosis
11. Pregnancy and women with child bearing potential without negative pregnancy test
12. Rupture not confirmed by CT or intra-operatively (impending ruptures are excluded)
13. RAAA requiring repair of the renal arteries or the proximal aorta

    * thoracoabdominal aneurysms requiring immediate repair
    * damaged renal arteries during emergency clamping requiring repair

Note:

* temporary clamping above the renal arteries (max 30 min total clamping time above the renal arteries) does not lead to exclusion
* ligation of the left renal vein does not lead to exclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-02-18 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2019-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harri Hakovirta, MD, Principal Investigator — Turku University Hospital; Maarit Venermo, MD, Principal Investigator — Helsinki University Central Hospital
Locations (9):
- Tartu University Hospital, Tartu, Estonia
- Finland (6):
  - Helsinki University Hospital, Helsinki
  - Central Finland Central Hospital, Jyväskylä
  - South Karelia Central Hospital, Lappeenranta
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kauno klinikos, Kaunas
  - Vilnius University Hospital Santaros klinikos, Vilnius

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hakovirta H, Jalkanen J, Saimanen E, Kukkonen T, Romsi P, Suominen V, Vikatmaa L, Valtonen M, Karvonen MK, Venermo M; INFORAAA Study Group. Induction of CD73 prevents death after emergency open aortic surgery for a ruptured abdominal aortic aneurysm: a randomized, double-blind, placebo-controlled study. Sci Rep. 2022 Feb 3;12(1):1839. doi: 10.1038/s41598-022-05771-1. PMID 35115574

RESULTS

PARTICIPANT FLOW:
Groups:
- FP-1201-lyo 10 µg: FP-1201-lyo 10 µg (Interferon Beta-1a) will be administered once daily as an intravenous bolus injection for 6 days.
  Investigational product is lyophilisate for solution for injection which will be reconstituted in water for injection.
  Interferon Beta-1a: investigational drug.
- FP-1201-lyo Placebo: FP-1201-lyo Placebo will be administered once daily as an intravenous bolus injection for 6 days.
  Investigational placebo is lyophilisate for solution for injection which will be reconstituted in water for injection
  Placebo: placebo for investigational drug.
Period: 6-day Dosing
Arm/Group | FP-1201-lyo 10 µg | FP-1201-lyo Placebo
Started | 29 | 11
Completed | 22 | 8
Not Completed | 7 | 3
Not completed — Death | 4 | 1
Not completed — Adverse Event | 3 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Mid-term (Final) Follow-up at D90
Arm/Group | FP-1201-lyo 10 µg | FP-1201-lyo Placebo
Started | 25 (3 patients who discontinued study drug due to adverse events were also followed up.) | 10 (2 patients who did not receive 6 doses were also followed up.)
Completed | 22 | 9
Not Completed | 3 | 1
Not completed — Death | 3 | 1

BASELINE CHARACTERISTICS:
Population: A total of 40 subjects received at least 1 dose of study drug. 2 patients were excluded from Full Analysis Set for Efficacy (FAS-E) and Per Protocol Set (PPS) populations due to early deaths (within 36 hours from first dose of the study treatment). Therefore, FAS-E and PPS populations consisted of 38 patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | FP-1201-lyo 10 µg | FP-1201-lyo Placebo | Total
Number analyzed (Participants) | 27 | 11 | 38
Age, Customized [Count of Participants; unit: Participants]
  < 70 years | 7 | 3 | 10
  70-80 years | 14 | 6 | 20
  > 80 years | 6 | 2 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4
  Male | 23 | 11 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 27 | 11 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Finland | 23 | 8 | 31
  Lithuania | 3 | 1 | 4
  Estonia | 1 | 2 | 3
Baseline Height [Mean (Standard Deviation); unit: centimetres] | 172.3 (6.34) | 177.5 (7.59) | 173.8 (7.05)
Baseline Weight [Mean (Standard Deviation); unit: kilograms] | 82.0 (16.14) | 95.9 (21.21) | 86.0 (18.58)

OUTCOME MEASURES:

1. Primary Outcome: The Efficacy of FP-1201-lyo Compared to Placebo Concerning All Cause Mortality
Description: Number of fatalities
Time Frame: Day 30
Population: The Full Analysis Set for Efficacy (FAS-E) defined as all randomised patients who received study treatment, excluding the early deaths (within 36 hours from first dose of the study treatment).
Measure: Count of Participants; unit: Participants
Arm/Group | FP-1201-lyo 10 µg | FP-1201-lyo Placebo
Number analyzed (Participants) | 27 | 11
Participants | 6 | 2
Statistical Analysis 1: Comparison: FP-1201-lyo 10 µg vs FP-1201-lyo Placebo; Test type: Superiority; p = 0.78, Regression, Logistic — The threshold for statistical significance was p = 0.05; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.21 to 8.19]

2. Secondary Outcome: The Efficacy of FP-1201-lyo Compared to Placebo Concerning All Cause Mortality
Description: Number of fatalities
Time Frame: Day 90
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | FP-1201-lyo 10 µg | FP-1201-lyo Placebo
Number analyzed (Participants) | 27 | 11
Participants | 7 | 2
Statistical Analysis 1: Comparison: FP-1201-lyo 10 µg vs FP-1201-lyo Placebo; Test type: Superiority; p = 0.57, Regression, Logistic — The threshold for statistical significance was p = 0.05; Odds Ratio (OR) = 1.7, 95% CI 2-sided [0.28 to 10.52]

3. Secondary Outcome: The Efficacy of FP-1201-lyo Compared to Placebo Concerning Number of Ventilator Free Days (VFDs)
Description: Number of ventilator free days. VFDs to Day 30 were defined as the number of calendar days after initiating unassisted breathing (UAB) to Day 30 from first treatment, assuming that a patient survives at least 48 consecutive hours after initiating UAB. Patients who die without initiating UAB were assigned a VFD value of zero.
Time Frame: Day 30
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | FP-1201-lyo 10 µg | FP-1201-lyo Placebo
Number analyzed (Participants) | 27 | 11
days | 25.0 [0.0 to 30.0] | 29.0 [0.0 to 29.0]
Statistical Analysis 1: Comparison: FP-1201-lyo 10 µg vs FP-1201-lyo Placebo; Test type: Superiority; p = 0.08, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p = 0.05

4. Secondary Outcome: The Efficacy of FP-1201-lyo Compared to Placebo Concerning Number of Days Receiving Hemodialysis
Description: Number of days receiving hemodialysis. There were only few reported values other than zero.
Time Frame: Day 30 and Day 90
Population: The Full Analysis Set for Efficacy (FAS-E) defined as all randomised patients who received study treatment, excluding the early deaths (within 36 hours from first dose of the study treatment).
  The overall number of participants analyzed reflects the number of patients that had sufficient data to allow for calculation of the outcome measure.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | FP-1201-lyo 10 µg | FP-1201-lyo Placebo
Number analyzed (Participants) | 21 | 9
days
  Day 30 | 0.9 (4.15) | 0.0 (0.00)
  Day 90: number analyzed (Participants) | 20 | 9
  Day 90 | 0.6 (2.68) | 0.0 (0.00)

5. Secondary Outcome: The Efficacy of FP-1201-lyo Compared to Placebo Concerning Number of Organ Failure Free Days by Means of the Sequential Organ Failure Assessment (SOFA) Score
Description: Organ failure free days were defined as the number of days in the first 30 days after the first dose of study medication that the patient was alive and free of organ failure with a SOFA score of zero for the following six organ parameters: respiration, coagulation, liver, cardiovascular, central nervous system and renal function. It is graded from 0 to 4 according to the degree of dysfunction/ failure (higher scores indicate more severe organ failure). Patients who died without achieving a SOFA score of zero was assigned an organ failure free days value of zero.
  Note: the information for organ failure free days has been only collected when the patients have been in the Intensive Care Unit (ICU). As ICU free days have been reported in a separate variable, it was decided that presented information will be kept, without trying to conduct imputation.
Time Frame: Day 30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | FP-1201-lyo 10 µg | FP-1201-lyo Placebo
Number analyzed (Participants) | 27 | 11
days | 0.0 (0.00) | 0.0 (0.00)
Statistical Analysis 1: Comparison: FP-1201-lyo 10 µg vs FP-1201-lyo Placebo; Test type: Superiority; p > 0.999, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p = 0.05

6. Secondary Outcome: The Efficacy of FP-1201-lyo Compared to Placebo Concerning Prevalence of Abdominal Compartment Syndrome by Intra-abdominal Pressure (IAP)
Description: Intra-abdominal pressure values, which were routinely measured during ICU stay via urine bladder catheter.
Time Frame: Days 1 - 6, D9 and D13 during Intensive Care Unit (ICU) stay
Population: The Full Analysis Set for Efficacy (FAS-E) defined as all randomised patients who received study treatment, excluding the early deaths (within 36 hours from first dose of the study treatment). The number of participants analyzed reflects the number of patients that were alive and had sufficient data to allow for calculation of the outcome measure.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | FP-1201-lyo 10 µg | FP-1201-lyo Placebo
Number analyzed (Participants) | 19 | 9
mmHg
  Day 1 | 15.4 (12.37) | 10.3 (4.80)
  Day 2: number analyzed (Participants) | 19 | 8
  Day 2 | 12.2 (3.58) | 12.1 (6.01)
  Day 3: number analyzed (Participants) | 16 | 6
  Day 3 | 13.1 (4.62) | 10.3 (5.35)
  Day 4: number analyzed (Participants) | 12 | 5
  Day 4 | 11.4 (6.60) | 8.6 (5.32)
  Day 5: number analyzed (Participants) | 10 | 4
  Day 5 | 10.5 (3.14) | 12.5 (5.45)
  Day 6: number analyzed (Participants) | 8 | 1
  Day 6 | 11.4 (5.29) | 15.0 (0)
  Day 9: number analyzed (Participants) | 4 | 0
  Day 9 | 11.0 (5.48) |
  Day 13: number analyzed (Participants) | 6 | 0
  Day 13 | 10.8 (4.49) |

7. Secondary Outcome: The Efficacy of FP-1201-lyo Compared to Placebo Concerning Neutralizing Antibodies Against IFN Beta-1a (NAbs) in Whole Blood Samples
Description: IFN beta-1a neutralizing antibodies immune response. Blood samples for the NAbs assessments were collected at Day 0 pre-dose (baseline) and at Day 30.
Time Frame: Day 30
Population: At the Baseline Visit, 2 patients in the FP-1201-lyo treatment group and 1 patient in the placebo treatment group were not tested for anti-drug antibodies.
Measure: Count of Participants; unit: Participants
Arm/Group | FP-1201-lyo 10 µg | FP-1201-lyo Placebo
Number analyzed (Participants) | 25 | 10
Participants
  Baseline | 0 | 0
  Day 30: number analyzed (Participants) | 19 | 9
  Day 30 | 0 | 0

8. Secondary Outcome: The Efficacy of FP-1201-lyo Compared to Placebo Concerning Disability by Modified Ranking Scale (mRS).
Description: Scale gives the degree of disability or dependence in the daily activities. Single mRS value is applied for every patient based on patient or caregiver interview. The scale runs from 0-6, from perfect health without symptoms to death. Pre-operation Baseline Visit mRS value is collected for reference.
Time Frame: Day 90
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | FP-1201-lyo 10 µg | FP-1201-lyo Placebo
Number analyzed (Participants) | 27 | 11
Participants
  No symptoms - 0 | 5 | 2
  No significant disability - 1 | 5 | 5
  Slight disability - 2 | 3 | 1
  Moderate disability - 3 | 2 | 0
  Moderately severe disability - 4 | 3 | 0
  Severe disability - 5 | 2 | 1
  Death - 6 | 7 | 2
Statistical Analysis 1: Comparison: FP-1201-lyo 10 µg vs FP-1201-lyo Placebo; Test type: Superiority; p = 0.3620, Mantel Haenszel — The threshold for statistical significance was p = 0.05; Exact Mantel-Haenszel Chi-Square Test

9. Secondary Outcome: Safety Parameters of Clinically Significant Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events, Vital Signs and Clinical Laboratory Parameters
Description: Number of TEAEs from vital signs data, laboratory data, physical examinations and spontaneous reporting when conscious.
Time Frame: Day 0 to Day 30
Population: The Full Analysis Set for Safety (FAS-S) consisted of all randomised patients receiving study treatment and comprised the analysis set on which the evaluation of safety is based.
Measure: Number; unit: Events
Arm/Group | FP-1201-lyo 10 µg | FP-1201-lyo Placebo
Number analyzed (Participants) | 29 | 11
Events
  Product-related TEAEs | 17 | 1
  Severe TEAEs | 28 | 2
  Serious TEAEs | 26 | 5
  TEAEs Leading to Study Product Discontinuation | 7 | 1
  TEAEs Leading to Death | 7 | 1

10. Secondary Outcome: Pharmacoeconomic Information of Length of ICU Stay, Length of Hospital Stay, Length of Stay at Another Health Care Facility, Length of Hemodialysis Needed, Ventilation Free Days
Description: Economic measurement:
  * Length of ICU stay, in terms of ICU free days at D30
  * Length of hospital stay, in terms of hospital free days at D90
  * Length of stay at another health care facility at D90
  * The number of days on hemodialysis at D30 and at D90
  * The number of organ failure free days at D30
  * The number of ventilation free days at D30
Time Frame: Day 30 or Day 90
Population: The Full Analysis Set for Efficacy (FAS-E). As the study was discontinued, analyses were performed on the available data gathered thus far.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | FP-1201-lyo 10 µg | FP-1201-lyo Placebo
Number analyzed (Participants) | 27 | 11
days
  ICU free days at Day 30 | 16.8 (12.39) | 21.9 (11.06)
  Days in hospital at Day 90: number analyzed (Participants) | 20 | 9
  Days in hospital at Day 90 | 18.1 (9.84) | 13.8 (9.97)
  Days in another facility at Day 90: number analyzed (Participants) | 15 | 8
  Days in another facility at Day 90 | 11.8 (23.79) | 7.0 (19.80)
  Days on hemodialysis at Day 30: number analyzed (Participants) | 21 | 9
  Days on hemodialysis at Day 30 | 0.9 (4.15) | 0.0 (0.00)
  Days on hemodialysis at Day 90: number analyzed (Participants) | 20 | 9
  Days on hemodialysis at Day 90 | 0.6 (2.68) | 0.0 (0.00)
  Organ failure free days at Day 30 | 0.0 (0.00) | 0.0 (0.00)
  Ventilation free days at Day 30 | 20.6 (10.62) | 25.1 (8.85)

11. Other Pre Specified Outcome: Myxovirus Resistant Protein A (MxA) Concentration in Whole Blood Samples as Pharmacodynamic Marker
Description: Concentration of Myxovirus Resistant Protein A (MxA)
Time Frame: Day 0 up to Day 13
Population: The Full Analysis Set for Efficacy (FAS-E) defined as all randomised patients who received study treatment, excluding the early deaths (within 36 hours from first dose of the study treatment). The overall number of participants analyzed reflects the number of patients that were alive and had data to allow for calculation of the outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | FP-1201-lyo 10 µg | FP-1201-lyo Placebo
Number analyzed (Participants) | 27 | 11
ng/mL
  Baseline | 3.5 [2.4 to 5.1] | 6.0 [3.3 to 11.0]
  Day 1 | 15.0 [10.2 to 22.1] | 5.1 [2.8 to 9.3]
  Day 2: number analyzed (Participants) | 27 | 10
  Day 2 | 19.8 [13.5 to 29.1] | 3.8 [2.1 to 7.0]
  Day 3: number analyzed (Participants) | 25 | 10
  Day 3 | 21.2 [14.3 to 31.4] | 3.3 [1.8 to 6.2]
  Day 4: number analyzed (Participants) | 23 | 9
  Day 4 | 36.4 [24.4 to 54.2] | 4.1 [2.2 to 7.7]
  Day 5: number analyzed (Participants) | 22 | 9
  Day 5 | 48.3 [32.3 to 72.3] | 3.1 [1.6 to 5.8]
  Day 6: number analyzed (Participants) | 23 | 8
  Day 6 | 50.4 [33.9 to 75.1] | 3.6 [1.9 to 6.8]
  Day 9: number analyzed (Participants) | 20 | 6
  Day 9 | 14.3 [9.5 to 21.5] | 4.8 [2.4 to 9.7]
  Day 13: number analyzed (Participants) | 17 | 3
  Day 13 | 3.9 [2.5 to 5.9] | 8.7 [3.7 to 20.7]
Statistical Analysis 1: Comparison: FP-1201-lyo 10 µg vs FP-1201-lyo Placebo; The lower limit of quantification (LLOQ) is equal 5 ng/ml. Values below the LLOQ were set to LLOQ/2 = 2.5 ng/ml. Values over the upper limit of quantitation (ULOQ) were set to 320 ng/ml; Test type: Superiority; p < .0001, ANOVA — Day 2, Day 3, Day 4, Day 5, and Day 6; Repeated measures ANOVA
Statistical Analysis 2: Comparison: FP-1201-lyo 10 µg vs FP-1201-lyo Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.13, ANOVA — Baseline visit; Repeated measures ANOVA
Statistical Analysis 3: Comparison: FP-1201-lyo 10 µg vs FP-1201-lyo Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.0035, ANOVA — Day 1; Repeated measures ANOVA
Statistical Analysis 4: Comparison: FP-1201-lyo 10 µg vs FP-1201-lyo Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.009, ANOVA — Day 9; Repeated measures ANOVA
Statistical Analysis 5: Comparison: FP-1201-lyo 10 µg vs FP-1201-lyo Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.10, ANOVA — Day 13; Repeated measures ANOVA

12. Other Pre Specified Outcome: Tentative Disease Specific Marker Cluster of Differentiation 73 (CD73, Ecto-5'-Nucleotidase Enzyme) Concentration in Serum Samples
Description: CD73 (ecto-5'-nucleotidase enzyme) concentration
Time Frame: Day 0 up to Day 13
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | FP-1201-lyo 10 µg | FP-1201-lyo Placebo
Number analyzed (Participants) | 27 | 11
ng/mL
  Baseline | 2.1 [1.8 to 2.5] | 2.2 [1.7 to 2.9]
  Day 1 | 2.0 [1.7 to 2.4] | 2.2 [1.6 to 2.8]
  Day 2: number analyzed (Participants) | 27 | 9
  Day 2 | 2.2 [1.8 to 2.6] | 2.2 [1.7 to 3.0]
  Day 3: number analyzed (Participants) | 25 | 10
  Day 3 | 2.0 [1.7 to 2.4] | 2.3 [1.7 to 3.1]
  Day 4: number analyzed (Participants) | 24 | 9
  Day 4 | 2.3 [1.9 to 2.8] | 2.6 [1.9 to 3.5]
  Day 5: number analyzed (Participants) | 23 | 9
  Day 5 | 3.0 [2.4 to 3.6] | 3.5 [2.6 to 4.8]
  Day 6: number analyzed (Participants) | 23 | 8
  Day 6 | 3.8 [3.2 to 4.6] | 3.8 [2.7 to 5.2]
  Day 9: number analyzed (Participants) | 20 | 6
  Day 9 | 3.9 [3.2 to 4.8] | 3.8 [2.6 to 5.4]
  Day 13: number analyzed (Participants) | 17 | 3
  Day 13 | 2.9 [2.3 to 3.6] | 2.7 [1.7 to 4.3]
Statistical Analysis 1: Comparison: FP-1201-lyo 10 µg vs FP-1201-lyo Placebo; Patients with an observation below the lower limit of quantification (LLOQ) value at baseline for CD73 were set to have the LLOQ value (LLOQ = 4 ng/ml) at baseline for subgroup determination purposes (2-fold increase in CD73 from baseline). Values below the LLOQ were set to LLOQ/2 = 2 ng/mL; Test type: Superiority; p = 0.66, ANOVA — The threshold for statistical significance was p = 0.05; Repeated measures ANOVA

13. Other Pre Specified Outcome: Tentative Disease Specific, Potential Inflammatory Marker - Interleukin 6 (IL-6) in Serum Samples
Description: IL-6 concentration.
Time Frame: Day 0 up to Day 13
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | FP-1201-lyo 10 µg | FP-1201-lyo Placebo
Number analyzed (Participants) | 27 | 11
pg/mL
  Baseline | 328.9 [223.8 to 483.3] | 378.9 [207.3 to 692.6]
  Day 1 | 493.1 [335.5 to 724.5] | 460.2 [251.8 to 841.0]
  Day 3: number analyzed (Participants) | 25 | 10
  Day 3 | 181.4 [122.0 to 270.0] | 130.7 [69.8 to 244.8]
  Day 6: number analyzed (Participants) | 22 | 8
  Day 6 | 164.1 [108.1 to 249.2] | 79.1 [39.8 to 157.1]
  Day 9: number analyzed (Participants) | 20 | 6
  Day 9 | 107.9 [69.9 to 166.5] | 74.5 [34.4 to 161.5]
Statistical Analysis 1: Comparison: FP-1201-lyo 10 µg vs FP-1201-lyo Placebo; Observations of zero were imputed as 1 pg/ml before logarithmic transformation; Test type: Superiority; p = 0.3, ANOVA — The threshold for statistical significance was p = 0.05; Repeated measures ANOVA

14. Other Pre Specified Outcome: Tentative Disease Specific, Potential Inflammatory Marker - Hepatocyte Growth Factor [HGF]) in Serum Samples
Description: HGF concentration.
Time Frame: Day 0 up to Day 13
Population: Data were not collected or analyzed due to the small groups and interference of corticosteroids it was not meaningful to perform the analyzes.
Arm/Group | FP-1201-lyo 10 µg | FP-1201-lyo Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The Adverse Event (AE) reporting period was up to study D30. In accordance with the protocol, the investigators reported AEs occurring after D30 only if the investigator considered a causal relationship with the study drug. All deaths were reported as SAEs throughout the study, up until D90.
Description: The "Serious Adverse Event" list and the "Other (Not including Serious) Adverse Event" list present all reported Treatment Emergent Adverse Events (defined as an AE that begins or that worsens in severity after at least one dose of study drug). In 3 study subjects a non-treatment emergent SAE began before first dose of the study drug (included in mortality numbers because these SAEs led to death)
Arm/Group | FP-1201-lyo 10 µg | FP-1201-lyo Placebo
All-Cause Mortality (participants affected / at risk) | 7/29 | 2/11
Serious Adverse Events (participants affected / at risk) | 13/29 | 3/11
Other Adverse Events (participants affected / at risk) | 27/29 | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FP-1201-lyo 10 µg (N=29) | FP-1201-lyo Placebo (N=11)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 3 (3) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 3 (3) | 0 (0)
Condition aggravated (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 4 (4) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Paraplegia (Nervous system disorders) | 1 (1) | 0 (0)
Spinal epidural haematoma (Nervous system disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FP-1201-lyo 10 µg (N=29) | FP-1201-lyo Placebo (N=11)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 5 (5) | 3 (4)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia paroxysmal (Cardiac disorders) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 6 (6) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 2 (2) | 0 (0)
Candida infection (Infections and infestations) | 2 (2) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 2 (2) | 0 (0)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Periprocedural myocardial infarction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural constipation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural oedema (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative delirium (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound secretion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood calcium decreased (Investigations) | 1 (1) | 0 (0)
Blood creatine increased (Investigations) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 2 (2) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Blood sodium increased (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 3 (3) | 1 (1)
Haemoglobin decreased (Investigations) | 4 (4) | 1 (1)
Hepatic enzyme increased (Investigations) | 3 (3) | 0 (0)
Inflammatory marker increased (Investigations) | 1 (1) | 0 (0)
Intra-abdominal pressure increased (Investigations) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 2 (2) | 1 (1)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0)
Urine output decreased (Investigations) | 2 (2) | 0 (0)
White blood cell count increased (Investigations) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Akathisia (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Confusional state (Psychiatric disorders) | 4 (4) | 2 (2)
Delirium (Psychiatric disorders) | 2 (2) | 1 (1)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Embolism arterial (Vascular disorders) | 0 (0) | 1 (2)
Hypertension (Vascular disorders) | 4 (4) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was prematurely stopped and due to this the planned statistical power for the primary comparisons was not reached.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-04-16): https://cdn.clinicaltrials.gov/large-docs/01/NCT03119701/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/01/NCT03119701/SAP_001.pdf